CLINICAL TRIAL: NCT00003741
Title: HeFi-1 Antibody Therapy in Ki-1 and Hodgkin's Lymphomas, a Phase I Study
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Refractory Anaplastic Large Cell Lymphoma or Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: BIDMC-97127; CDR0000066859 (Registry Identifier: PDQ (Physician Data Query)); NEDH-97127; NCI-870; NCI-V99-1515
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2005-03

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; anaplastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic

INTERVENTIONS:
Biological: monoclonal antibody HeFi-1

SUMMARY:
RATIONALE: Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of monoclonal antibody therapy in treating patients with refractory anaplastic large cell lymphoma or Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and tolerability of multiple doses of monoclonal antibody HeFi-1 in patients with CD30+ anaplastic large cell lymphoma or Hodgkin's lymphoma.
* Determine the pharmacokinetics of this drug in this patient population.
* Evaluate the efficacy, in terms of correlating immunologic parameters and immunogenicity, of this drug in these patients.

OUTLINE: This is an open-label, dose-escalation study.

Patients receive monoclonal antibody HeFi-1 IV over 30 minutes 3 times a week for 2 weeks. Treatment may continue for 2 additional weeks in the absence of anti-HeFi-1 response. Responding patients may continue treatment at monthly intervals for one year.

Cohorts of 3-4 patients receive escalating doses of monoclonal antibody HeFi-1 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 4 patients experience dose-limiting toxicity.

Patients are followed monthly.

PROJECTED ACCRUAL: A total of 9 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed CD30+ anaplastic large cell lymphoma (ALCL) or Hodgkin's lymphoma

  * At least 50% of malignant cells must react with HeFi-1
  * HIV positive or HIV negative
* Measurable disease
* No symptomatic CNS disease
* Must have failed or be ineligible for standard chemotherapy regimen

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* More than 2 months

Hematopoietic:

* Not specified

Hepatic:

* No significant hepatic disease
* Bilirubin no greater than 2 mg/dL

Renal:

* No significant renal disease
* Creatinine no greater than 3 mg/dL

Cardiovascular:

* No significant cardiovascular disease

Pulmonary:

* No significant pulmonary disease

Other:

* No significant endocrine, rheumatologic, or allergic disease
* No active clinical disease caused by cytomegalovirus (CMV), herpes simplex virus (HSV) I, HSV II, hepatitis B, or tuberculosis
* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior murine antibody therapy

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy to measurable disease

Surgery:

* Not specified

Other

* At least 4 weeks since prior cytotoxic therapy to measurable disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-02; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Koon, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States